CLINICAL TRIAL: NCT04229836
Title: An International, Multicentre, Open- Label, Interventional Phase IV Clinical Study to Investigate the Efficacy and Safety of Tildrakizumab 100 mg in Patients With Moderate- Severe Chronic Plaque Psoriasis and Its Impact on Their Quality of Life (TRIBUTE)
Brief Title: Efficacy and Safety of Tildrakizumab 100 Milligrams (mg) in Participants With Moderate-Severe Chronic Plaque Psoriasis and Its Impact on Their Quality of Life (TRIBUTE)
Acronym: TRIBUTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-14745-42
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Plaque Psoriasis
Keywords: Tildrakizumab; Moderate-to-Severe Chronic Plaque Psoriasis; Quality of Life (QoL)
MeSH Terms: interventions — tildrakizumab; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tildrakizumab (Experimental): Participants will receive subcutaneous (SC) injection of tildrakizumab 100 milligrams (mg).
  Interventions: Drug: Tildrakizumab 100 mg Solution for Injection

INTERVENTIONS:
Drug: Tildrakizumab 100 mg Solution for Injection — Participants will be treated with tildrakizumab 100 mg.

SUMMARY:
The main aim of the study is to evaluate the efficacy, safety and impact on the health-related quality of life (HRQoL) in participants with moderate-to-severe chronic plaque psoriasis who are treated with tildrakizumab 100 milligrams (mg).

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written and dated informed consent given before any study related activity is performed
* Participants with a diagnosis of moderate to severe plaque psoriasis
* Participants eligible for systemic biologic treatment as assessed by the investigator or having had a primary/secondary failure to treatment with one or more anti-Tumor Necrosis Factor (TNF) biologic agents for psoriasis

Exclusion Criteria:

* Unable to comply with the requirements of the study or who in the opinion of the study physician should not participate in the study
* Participants meeting any of the exclusion criteria specified in the summary of product characteristics (SmPC) of Ilumetri®
* Women currently pregnant, or intend to become pregnant or breastfeeding. Unwillingness/inability for the participants (women or men) to use appropriate measures of contraception (if necessary)
* Other forms of psoriasis than chronic plaque-type
* Current severe and/or uncontrolled psoriatic arthritis (PsA), or participants with PsA that is currently receiving systemic treatment
* Drug-induced psoriasis at the Screening Visit
* Concurrent malignancy, current relevant autoimmune diseases other than psoriasis
* Participants with severe renal impairment, haematological abnormality and abnormal liver enzymes at the screening visit
* Active infection disease or history of recurrent infection
* Active or latent tuberculosis (TB) at Screening visit
* Positive test for human immunodeficiency virus or any other immunosuppressive disease
* Participants with exposure to psoriasis systemic investigational drugs in the previous year
* Live vaccination within 4 weeks prior to the Baseline Visit
* Participants who intend to use any concomitant medication with immunomodulating or systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Absolute Psoriasis Area and Severity Index (PASI) Score at Week 24 | Week 24
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease).
Change from Baseline in the Absolute Psoriasis Area and Severity Index (PASI) Score at Week 24 | Baseline (Day 1) and Week 24
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease). Change from baseline will be calculated by subtracting post-dose value baseline value.
Absolute Dermatology Life Quality Index (DLQI) Score at Week 24 | Week 24
  DLQI is a questionnaire which is to evaluate the impact on participant's quality of life due to psoriasis. It is composed of ten items related to symptoms, feelings, daily activities, leisure, working or studying activities, personal relationships and opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30.
Change from Baseline in the Absolute Dermatology Life Quality Index (DLQI) Score at Week 24 | Baseline (Day 1) and Week 24
  DLQI is a questionnaire which is to evaluate the impact on participant's quality of life due to psoriasis. It is composed of ten items related to symptoms, feelings, daily activities, leisure, working or studying activities, personal relationships and opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30. Change from baseline will be calculated by subtracting post-dose value baseline value.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Absolute Dermatology Life Quality Index (DLQI) Scores Between 0-1 at Week 24 | Week 24
  DLQI is a questionnaire which is to evaluate the impact on participant's quality of life due to psoriasis. It is composed of ten items related to symptoms, feelings, daily activities, leisure, working or studying activities, personal relationships and opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30.
Percentage of Participants Achieving Absolute Dermatology Quality of Life Index Relevant (DLQI-R) Score Between 0-1 at Week 24. | Week 24
  DLQI-R is a scoring modification for the DLQI to better evaluate not relevant responses on the DLQI that could lead to underestimation of the impact on quality of life. The DLQI-R scoring modification involves multiplying the original DLQI score by a conversion factor that increases with the number of not relevant responses.
Absolute Dermatology Life Quality Index (DLQI) Score | Baseline (Day 1), Week 4, 16, 24
  DLQI is a questionnaire which is to evaluate the impact on participant's quality of life due to psoriasis. It is composed of ten items related to symptoms, feelings, daily activities, leisure, working or studying activities, personal relationships and opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30.
Change from Baseline in the Absolute Dermatology Life Quality Index (DLQI) Score | Baseline (Day 1), Week 4, 16, 24
  DLQI is a questionnaire which is to evaluate the impact on participant's quality of life due to psoriasis. It is composed of ten items related to symptoms, feelings, daily activities, leisure, working or studying activities, personal relationships and opinions about dermatological treatment. Each item is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30. Change from baseline will be calculated by subtracting post-dose value baseline value.
Absolute Dermatology Quality of Life Index Relevant (DLQI-R) Score | Baseline (Day 1), Week 4, 16, 24
  DLQI-R is a scoring modification for the DLQI to better evaluate not relevant responses on the DLQI that could lead to underestimation of the impact on quality of life. The DLQI-R scoring modification involves multiplying the original DLQI score by a conversion factor that increases with the number of not relevant responses.
Change from Baseline in the Absolute Dermatology Quality of Life Index Relevant (DLQI-R) Score | Baseline (Day 1), Week 4, 16, 24
  DLQI-R is a scoring modification for the DLQI to better evaluate not relevant responses on the DLQI that could lead to underestimation of the impact on quality of life. The DLQI-R scoring modification involves multiplying the original DLQI score by a conversion factor that increases with the number of not relevant responses. Change from baseline will be calculated by subtracting post-dose value baseline value.
Percentage of Participants Achieving Absolute Psoriasis Area and Severity Index (PASI) Score of 5, 3, and 1 | Baseline (Day 1), Week 4, 16, 24
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease).
Absolute Psoriasis Area and Severity Index (PASI) Score | Baseline (Day 1), Week 4, 16, 24
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease).
Change from Baseline in the Absolute Psoriasis Area and Severity Index (PASI) Score | Baseline (Day 1), Week 4, 16, 24
  PASI is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and scaling on a scale range from 0 (no symptoms) to 4 (very marked), together with the percentage (%) of the area affected, rated on a scale from 0 (0%) to 6 (90-100%). PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 (no psoriasis) to 72 (the most severe disease). Change from baseline will be calculated by subtracting post-dose value baseline value.
Absolute Physician Global Assessment (PGA) Score | Baseline (Day 1), Week 4, 16, 24
  The PGA used to assess the overall severity of the psoriasis lesions at the time of evaluation. Overall lesions will be graded for erythema, induration, and scale based on 6-point scale ranging from 0 (clear) to 5 (severe). The sum of 3 scales will be divided by 3 to obtain final PGA score.
Change from Baseline in the Absolute Physician Global Assessment (PGA) Score | Baseline (Day 1), Week 4, 16, 24
  The PGA used to assess the overall severity of the psoriasis lesions at the time of evaluation. Overall lesions will be graded for erythema, induration, and scale based on 6-point scale ranging from 0 (clear) to 5 (severe). The sum of 3 scales will be divided by 3 to obtain final PGA score. Change from baseline will be calculated by subtracting post-dose value baseline value.
Percentage of Participants Achieving Physician Global Assessment (PGA) Score of 0 or 1 with At Least a 2-Grade Reduction from Baseline | Baseline (Day 1), Week 4, 16, 24
  The PGA used to assess the overall severity of the psoriasis lesions at the time of evaluation. Overall lesions will be graded for erythema, induration, and scale based on 6-point scale ranging from 0 (clear) to 5 (severe). The sum of 3 scales will be divided by 3 to obtain final PGA score.
Absolute Body Surface Area (BSA) Score | Baseline (Day 1), Week 4, 16, 24
  BSA is a numerical score used to measure the total area of the body affected by psoriasis. The palm method will be applied: the participant's palm, including the five digits is used as a reference (representing approximately 1% of the total body surface area) and is used to repeatedly cover the lesions on the body. The investigator totals the number of palms required and then estimates the percentage (%) in each of the four body regions: head (including scalp) and neck (10%); upper extremities (20%); trunk (30%); and lower extremities (40%).
Change from Baseline in the Absolute Body Surface Area (BSA) Score | Baseline (Day 1), Week 4, 16, 24
  BSA is a numerical score used to measure the total area of the body affected by psoriasis. The palm method will be applied: the participant's palm, including the five digits is used as a reference (representing approximately 1% of the total body surface area) and is used to repeatedly cover the lesions on the body. The Investigator totals the number of palms required and then estimates the percentage (%) in each of the four body regions: head (including scalp) and neck (10%); upper extremities (20%); trunk (30%); and lower extremities (40%). Change from baseline will be calculated by subtracting post-dose value baseline value.
Absolute Pruritus-Numerical Rating Scale (NRS) Score | Baseline (Day 1), Week 4, 16, 24
  Pruritus is assessed by ticking the number on a 11 points scale, going from 0 - no pruritus, to 10 - worst imaginable pruritus. Higher scores depict worst pain.
Change from Baseline in the Absolute Pruritus-Numerical Rating Scale (NRS) Score | Baseline (Day 1), Week 4, 16, 24
  Pruritus is assessed by ticking the number on a 11 points scale, going from 0 - no pruritus, to 10 - worst imaginable pruritus. Change from baseline will be calculated by subtracting post-dose value baseline value.
Absolute Pain-Numerical Rating Scale (NRS) Score | Baseline (Day 1), Week 4, 16, 24
  The pain-NRS is an 11-point ordinal scale assessing pain, from 0 (no pain) to 10 (worst imaginable pain). Higher scores depict worst pain.
Change from Baseline in the Absolute Pain-Numerical Rating Scale (NRS) Score | Baseline (Day 1), Week 4, 16, 24
  The pain-NRS is an 11-point ordinal scale assessing pain, from 0 (no pain) to 10 (worst imaginable pain). Higher scores depict worst pain. Change from baseline will be calculated by subtracting post-dose value baseline value.
Absolute Scaling-Numerical Rating Scale (NRS) Score | Baseline (Day 1), Week 4, 16, 24
  The scaling-NRS is an 11-point ordinal scale assessing scaling, from 0 (no pain) to 10 (worst imaginable pain). Higher scores depict worst pain.
Change from Baseline in the Absolute Scaling-Numerical Rating Scale (NRS) Score | Baseline (Day 1), Week 4, 16, 24
  The scaling-NRS is an 11-point ordinal scale assessing scaling, from 0 (no pain) to 10 (worst imaginable pain). Higher scores depict worst pain. Change from baseline will be calculated by subtracting post-dose value baseline value.
Absolute Skindex-16 Questionnaire Score at Week 24 | Week 24
  Skindex is the best dermatological instruments to measure dermatology-specific health-related quality of life (HRQoL). The 16-item Skindex questionnaire is divided into three domains: questions related to the participant's symptoms (1- 4), emotions (5 -11), and functioning (12-16). Each question asks the participant to quantify how much a specific aspect of their skin condition bothered them in the week prior to administration of the Skindex-16. The questions are answered on a scale from 0 (never bothered) to 6 (always bothered) with a total possible score ranging from 0 (best HRQoL) to 96 (worst HRQoL). Each item is then transformed to a linear scale from 0 to 100.
Change from Baseline in the Absolute Skindex-16 Questionnaire Score at Week 24 | Baseline (Day 1) and Week 24
  Skindex is the best dermatological instruments to measure dermatology-specific health-related quality of life (HRQoL). The 16-item Skindex questionnaire is divided into three domains: questions related to the participant's symptoms (1-4), emotions (5-11), and functioning (12-16). Each question asks the participant to quantify how much a specific aspect of their skin condition bothered them in the week prior to administration of the Skindex-16. The questions are answered on a scale from 0 (never bothered) to 6 (always bothered) with a total possible score ranging from 0 (best HRQoL) to 96 (worst HRQoL). Each item is then transformed to a linear scale from 0 to 100. Change from baseline will be calculated by subtracting post-dose value baseline value.
Absolute Medical Outcome Study (MOS) Sleep Score at Baseline and Week 24 | Baseline (Day 1) and Week 24
  The MOS-Sleep includes 12 items assessing sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache. Subscales are standardised to yield scores from 0 to 100, with the exception of sleep quantity. Higher scores on the MOS sleep reflects more of the attribute indicated by the subscale name.
Change from Baseline in the Absolute Medical Outcome Study (MOS) Sleep Score at Baseline and Week 24 | Baseline (Day 1) and Week 24
  The MOS-Sleep includes 12 items assessing sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache. Subscales are standardised to yield scores from 0 to 100, with the exception of sleep quantity. Higher scores on the MOS sleep reflects more of the attribute indicated by the subscale name. Change from baseline will be calculated by subtracting post-dose value baseline value.
Absolute Work Productivity and Activity Impairment (WPAI) Score at Week 24 | Week 24
  The WPAI questionnaire is an instrument to measure impairments in both paid work and unpaid work. The WPAI questionnaire consists of 6 questions that are used to assess: 1-employment status (yes/no), 2- work time missed due to Psoriasis (hours), 3-work time missed due to other reasons (hours), 4-actual work time (hours), 5-the impact of Psoriasis on work productivity while at work (0:10 point scale), and 6-the impact of Psoriasis on activities outside of work (0:10 point scale) for the 7 days prior to questionnaire completion. Four scores are derived from the questions: percent absenteeism (work time missed), percent presenteeism (impairment at work), percent work productivity loss (overall work impairment due to absenteeism and presenteeism), and percent activity impairment (activities performed outside of work). Higher scores indicate a higher level of impairment.
Change from Baseline in the Absolute Work Productivity and Activity Impairment (WPAI) Score at Week 24 | Baseline (Day 1) and Week 24
  The WPAI questionnaire is an instrument to measure impairments in both paid work and unpaid work. The WPAI questionnaire consists of 6 questions that are used to assess: 1-employment status (yes/no), 2- work time missed due to Psoriasis (hours), 3-work time missed due to other reasons (hours), 4-actual work time (hours), 5-the impact of Psoriasis on work productivity while at work (0:10 point scale), and 6-the impact of Psoriasis on activities outside of work (0:10 point scale) for the 7 days prior to questionnaire completion. Four scores are derived from the questions: percent absenteeism (work time missed), percent presenteeism (impairment at work), percent work productivity loss (overall work impairment due to absenteeism and presenteeism), and percent activity impairment (activities performed outside of work). Higher scores indicate a higher level of impairment. Change from baseline will be calculated by subtracting post-dose value baseline value.
Absolute Treatment Satisfaction Questionnaire for Medication (TSQM) Score at Week 24 | Week 24
  The TSQM is a 14-item self-reported generic instrument designed to measure participant satisfaction with medication treatment. The 4 scales of the TSQM include the Effectiveness subscale, the Side Effects subscale (items 4-8), the Convenience subscale (items 9-11), and the Global Satisfaction subscale (items 12-14). The last subscale is regarded both in concept and in research as a superordinate, second-order global factor encompassing the other 3 more specific domains of medication experiences. Responses are obtained on a 5-point or a 7-point Likert scale (range, 1 extremely dissatisfied'' to 7 extremely satisfied'') for all but 1 item that has a yes-no response option. The subscale scores are transformed into scores ranging from 0 to 100, with higher scores representing higher satisfaction on that domain. Regarding the Side Effects subscale, when the participant answers no'' to experiencing side effects (item 4), this subscale is scored as 100.
Percentage of Participants Achieving a Score Greater Than or Equal to (>=) 1 in the Absolute Patient Benefit Index (PBI) Score at Week 24. | Week 24
  This is a questionnaire of 23 items on participant-relevant therapy needs and benefits. The first part of the instrument, the Participant Needs Questionnaire (PNQ), is filled in by the participant before therapy. A five- step Likert scale (0 = not important at all to 4 = very important) records the individual relevance of the different items to the participant. The second part, the Participant Benefit Questionnaire (PBQ), is filled in by the participants during or after therapy. It comprises the same items as the PNQ, but in contrast, the participants evaluate the extent to which the treatment needs have been fulfilled by therapy (scaled from 0 = treatment did not help at all to 4 = treatment helped a lot). In addition, the Likert scale contains the option does not apply to me in the PNQ and the option did not apply to me in the PBQ. This questionnaire score ranges from 0 = no benefit to 4 = maximal benefit. A PBI value of >=1 is considered as relevant benefit.
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Baseline (Day 1) up to Week 28
  An Adverse Event (AE) will be considered as TEAE if it was not present prior to the first dose of the study drug or was present prior to the first dose of study drug, but increased in severity during the treatment period.
Absolute High-sensitivity C-Reactive Protein (hs-CRP) at Week 24 | Week 24
  The hs-CRP will be assessed as safety serum biochemistry parameters.
Change from Baseline in the Absolute High-sensitivity C-Reactive Protein (hs-CRP) at Week 24 | Baseline (Day 1) and Week 24
  The hs-CRP will be assessed as safety serum biochemistry parameters. Change from baseline will be calculated by subtracting post-dose value baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, SAS
Locations (39):
- Italy (19):
  - Investigator Site 9, Ancona
  - Investigator Site 11, Arezzo
  - Investigator Site 7, Cagliari
  - Investigator Site 15, Catania
  - Investigator Site 14, Erice
  - Investigator Site 4, Genova
  - Investigator Site 6, L’Aquila
  - Investigator Site 12, Milan
  - Investigator Site 2, Modena
  - Investigator Site 13, Napoli
  - Investigator Site 10, Novara
  - Investigator Site 16, Parma
  - Investigator Site 18, Perugia
  - Investigator Site 19, Reggio Calabria
  - Investigator Site 17, Roma
  - Investigator Site 3, Roma
  - Investigator Site 5, Roma
  - Investigator Site 1, Rozzano (MI)
  - Investigator Site 8, Torino
- Spain (20):
  - Investigator Site 14, A Coruña
  - Investigator Site 18, Albacete
  - Investigator Site 12, Alicante
  - Investigator Site 20, Barcelona
  - Investigator Site 2, Barcelona
  - Investigator Site 3, Barcelona
  - Investigator Site 4, Barcelona
  - Investigator Site 16, Granada
  - Investigator Site 22, Granada
  - Investigator Site 1, Las Palmas
  - Investigator Site 19, Madrid
  - Investigator Site 21, Madrid
  - Investigator Site 6, Madrid
  - Investigator Site 7, Madrid
  - Investigator Site 8, Madrid
  - Investigator Site 9, Madrid
  - Investigator Site 13, Pontevedra
  - Investigator Site 11, Valencia
  - Investigator Site 17, Valencia
  - Investigator Site 15, Zaragoza